CLINICAL TRIAL: NCT06532565
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of GS-2121 as Monotherapy and in Combination in Adults With Advanced Solid Tumors
Brief Title: Study of GS-2121 Given Alone or in Combination in Adults With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-579-6764; 2024-511739-81 (Other: European Medicines Agency)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: GS-2121 Monotherapy Dose Escalation (Experimental): Participants will receive escalating doses of GS-2121 monotherapy until disease progression, or until the participant meets other study drug discontinuation criteria as specified in protocol.
  Interventions: Drug: GS-2121
- Part B: GS-2121 Monotherapy Dose Expansion (Experimental): Participants with selected indications will receive GS-2121 monotherapy at the recommended dose for expansion.
  Interventions: Drug: GS-2121
- Part C: Combination Dose Escalation of GS-2121 with Zimberelimab (Experimental): Participants will receive escalating doses of GS-2121 in combination with zimberelimab until disease progression, or until the participant meets other study drug discontinuation criteria as specified in protocol.
  Interventions: Drug: GS-2121; Drug: Zimberelimab
- Part D: Combination Dose Expansion of GS-2121 with Zimberelimab (Experimental): Participants with selected indications will receive GS-2121 at the recommended dose for expansion in combination with zimberelimab.
  Interventions: Drug: GS-2121; Drug: Zimberelimab

INTERVENTIONS:
Drug: GS-2121 — Tablet administered orally
Drug: Zimberelimab — Administered intravenously
  Other Names: GS-0122; AB122
  Arms: Part C: Combination Dose Escalation of GS-2121 with Zimberelimab; Part D: Combination Dose Expansion of GS-2121 with Zimberelimab

SUMMARY:
The main goal of this first-in-human (FIH) study is to learn about the safety and dosing of GS-2121 when given alone or in combination with zimberelimab (ZIM) in participants with advanced solid tumors.

The primary objectives of this study are:

* To assess the safety and tolerability of GS-2121 as monotherapy and GS-2121 in combination with zimberelimab in participants with advanced solid tumors.
* To identify the maximum tolerated dose (MTD) / maximum administered dose (MAD) and/or the recommended phase 2 dose (RP2D) of GS-2121 as monotherapy and in combination with zimberelimab in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants diagnosed with histologically or cytologically confirmed advanced solid tumors who have progressed despite standard therapy, are intolerant to standard therapy, or are ineligible for standard therapy.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Tissue requirements:

  1. Parts A-D: Pretreatment tumor tissue is required.
  2. Parts A and C backfill cohorts: Participants must agree to fresh pre- and on-treatment biopsies.
* Adequate organ function.

Key Exclusion Criteria:

* Positive serum pregnancy test or participant who is breastfeeding.
* Requirement for ongoing therapy with any prohibited medications.
* Any anti-cancer therapy, whether investigational or approved within protocol specified time prior to initiation of study including: major surgery (<4 weeks), experimental therapy (<21 days or <5 half-lives whichever is longer), approved immunotherapy or biologic therapy (<28 days), approved chemotherapy (<21 days or <42 days for mitomycin or nitrosoureas), approved targeted small molecule therapy (<14 days or <5 half-lives whichever is longer), hormonal therapy or other adjunctive therapy for cancers other than cancer under evaluation in this study (<14 days) or radiation therapy (<21 days).
* Any prior allogeneic tissue/solid organ transplantation, including allogeneic stem cell transplantation.
* Have not recovered (ie, returned to Grade 1 or baseline) from AEs due to a previously administered agent.
* Have known active central nervous system (CNS) metastases and/or leptomeningeal disease (LMD).
* Diagnosis of immunodeficiency, either primary or acquired.
* History of autoimmune disease or active autoimmune disease that has required systemic treatment within 2 years prior to the start of study treatment.
* Have an active second malignancy.
* Active and clinically relevant bacterial, fungal, or viral infection that is not controlled or requires systemic antibiotics, antifungals, or antivirals, respectively.
* History of pneumonitis requiring treatment with corticosteroids, interstitial lung disease, or severe radiation pneumonitis (excluding localized radiation pneumonitis).
* Ascites or pleural effusion that is symptomatic and/or requiring medical intervention.
* Have active hepatitis B virus (HBV) or hepatitis C virus (HCV), or HIV.
* Meet any of the following criteria for cardiac disease: Myocardial infarction or unstable angina pectoris within 6 months of enrollment. History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication). Mean QT interval corrected for heart rate using the Fridericia's formula (QTcF) ≥ 470 msec. New York Heart Association Class > III congestive heart failure or known left ventricular ejection fraction < 40%.
* Live vaccines within 28 days of initiation of study drug(s).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Parts A and B: Percentage of Participants with Adverse Events and Serious Adverse Events | First dose up to 90 days post last dose (up to approximately 118 weeks)
Parts A and B: Percentage of Participants with Laboratory Abnormalities | First dose up to 90 days post last dose (up to approximately 118 weeks)
Part A: Percentage of Participants with Dose-Limiting Toxicities (DLTs) During Dose Escalation | Day 1 up to Day 21
  DLTs are defined as any of the protocol-specified treatment-emergent adverse events (AEs) with onset within the DLT-evaluation period for the corresponding dose.
Parts C and D: Percentage of Participants with Adverse Events and Serious Adverse Events | First dose up to 90 days post last dose (up to approximately 118 weeks)
Parts C and D: Percentage of Participants with Laboratory Abnormalities | First dose up to 90 days post last dose (up to approximately 118 weeks)
Part C: Percentage of Participants with DLTs During Dose Escalation | Day 1 up to Day 21
  DLTs are defined as any of the protocol-specified treatment-emergent adverse events (AEs) with onset within the DLT-evaluation period for the corresponding dose.

SECONDARY OUTCOMES:
Parts A and B: Plasma Concentration of GS-2121 and Active Metabolite | Predose and postdose up to end of treatment (up to 105 weeks)
Parts A and B: PK Parameter: AUC0-24 of GS-2121 | Predose and postdose up to end of treatment (up to 105 weeks)
  AUC0-24 is defined as the partial area under the concentration of drug over time between time 0 and time 24 hours. PK parameters will be estimated as applicable, based on the availability of data.
Parts A and B: PK Parameter: Cmax of GS-2121 | Predose and postdose up to end of treatment (up to 105 weeks)
  Cmax is defined as the maximum observed drug concentration. PK parameters will be estimated as applicable, based on the availability of data.
Parts A and B: PK Parameter: Tmax of GS-2121 | Predose and postdose up to end of treatment (up to 105 weeks)
  Tmax is defined as the time to maximum observed drug concentration. PK parameters will be estimated as applicable, based on the availability of data.
Parts C and D: Plasma Concentration of GS-2121 and Active Metabolite | Predose and postdose up to end of treatment (up to 105 weeks)
Parts C and D: PK Parameter: AUC0-24 of GS-2121 | Predose and postdose up to end of treatment (up to 105 weeks)
  AUC0-24 is defined as the partial area under the concentration of drug over time between time 0 and time 24 hours. PK parameters will be estimated as applicable, based on the availability of data.
Parts C and D: PK Parameter: Cmax of GS-2121 | Predose and postdose up to end of treatment (up to 105 weeks)
  Cmax is defined as the maximum observed drug concentration. PK parameters will be estimated as applicable, based on the availability of data.
Parts C and D: PK Parameter: Tmax of GS-2121 | Predose and postdose up to end of treatment (up to 105 weeks)
  Tmax is defined as the time to maximum observed drug concentration. PK parameters will be estimated as applicable, based on the availability of data.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (4):
  - Stanford Cancer Center, Palo Alto, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - NEXT Oncology, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa
  - Princess Margaret Cancer Centre, Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06532565